CLINICAL TRIAL: NCT07406165
Title: ShotBlocker and Helfer Technique in the Management of Pain and Fear During Hormone Injection in Patients With Breast Cancer: A Randomized Controlled Trial
Brief Title: Nonpharmacological Management of Pain and Fear During Hormone Injection in Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha CENGİZ, Associate Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: INONU-BC-2026-01; 9222 (Other: Inonu University Health Sciences Scientific Research Ethics Committee)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Pain and Fear During Intramuscular Hormone Injections
Keywords: Breast cancer, Hormone therapy, Intramuscular injection, Injection pain, Injection fear
MeSH Terms: conditions — Breast Neoplasms; Pain; Iatrophobia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to three parallel groups: ShotBlocker, Helfer Skin Tap Technique, and Control. Each group will receive only its assigned intervention during the study period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ShotBlocker Group (Experimental): Shotblocker Group: The Shotblocker device will be positioned at the gluteal injection site using aseptic techniques immediately before the administration of hormonal medications. Standard intramuscular (IM) injection protocols will be followed while the device is in situ to mitigate injection-related pain.
  Interventions: Device: ShotBlocker device
- Helfer Skin Tap Technique Group (Active Comparator): Helfer Skin Tap Group: Rhythmic skin tapping will be performed at points near the gluteal injection site immediately before and during the procedure. Standard intramuscular (IM) injection of hormonal medications will be administered following the Helfer Skin Tap protocol to reduce procedural pain and muscle tension.
  Interventions: Procedure: This involves rhythmic, gentle tapping with the fingertips on the skin surrounding the gluteal injection site.
- Control Group (No Intervention): Control Group: Standard intramuscular (IM) injection of hormonal medications will be administered to participants in this group without any supportive technique. The procedure will follow routine clinical nursing protocols.

INTERVENTIONS:
Device: ShotBlocker device — Participants in this group will receive intramuscular (IM) injections of premenopausal or postmenopausal hormonal medications. Immediately prior to the procedure, the Shotblocker device (a plastic, butterfly-shaped tool with blunt contact points) will be applied to the gluteal muscle injection site following aseptic techniques. The device will be pressed firmly against the skin to saturate the sensory signals through the gate control mechanism. While the device is in place, the IM injection will be administered according to standard clinical protocols. The device will be removed once the injection is completed and the needle is withdrawn.
  Arms: ShotBlocker Group
Procedure: This involves rhythmic, gentle tapping with the fingertips on the skin surrounding the gluteal injection site. — Participants in this group will receive intramuscular (IM) injections of premenopausal or postmenopausal hormonal medications. Prior to and during the injection, the Helfer Skin Tap (HST) technique will be applied. This involves rhythmic, gentle tapping with the fingertips on the skin surrounding the gluteal injection site. The tapping starts just before the needle insertion and continues rhythmically to promote muscle relaxation and utilize the gate control theory of pain management. The IM injection will be administered according to standard clinical protocols while maintaining the rhythmic tapping.
  Arms: Helfer Skin Tap Technique Group

SUMMARY:
This randomized controlled study will compare the effects of the ShotBlocker device and the Helfer Skin Tap Technique on pain and fear during intramuscular hormone injections in premenopausal and postmenopausal breast cancer patients. Ninety-nine participants will be randomly assigned to three groups (ShotBlocker, Helfer, control). All injections will be administered by the same nurse using standardized procedures. Pain will be assessed with the Visual Analog Scale, and fear with the Injection Fear Scale. The study aims to identify effective nonpharmacological methods to enhance patient comfort, support treatment adherence, and improve nursing care quality.

DETAILED DESCRIPTION:
Objective This study aims to comparatively evaluate the effects of the ShotBlocker device and the Helfer Skin Tap Technique on pain and fear during intramuscular (IM) injection of premenopausal and postmenopausal hormone medications used in breast cancer patients. The study aims to increase patient comfort, support treatment compliance, and improve the quality of nursing care.

Type of Research This research will be conducted using a randomized controlled experimental design. Participants will be randomly assigned to three groups: the ShotBlocker group, the Helfer Skin Tap Technique group, and the control group.

Location and Time of the Study The study will be conducted in the oncology unit of Batman Training and Research Hospital between February and April 2026.

Participants/Sample The study population consists of premenopausal and postmenopausal breast cancer patients who apply to the hospital for hormone injection during the specified dates. Power analysis calculated a minimum of 93 patients; considering possible losses, a total of 99 patients is targeted. Participants will be distributed equally among the groups (ShotBlocker=33, Helfer=33, Control=33).

Method / Intervention ShotBlocker Group: The ShotBlocker device will be placed in the gluteal region prior to injection.

Helfer Skin Tap Technique Group: Points close to the injection site will be stimulated with rhythmic taps prior to injection.

Control Group: The standard IM injection protocol will be applied. All injections will be administered by the same nurse, using the same technique, in a standardized manner. Pain will be assessed using the Visual Analog Scale (VAS) after the injection, and fear will be assessed using the Injection Fear Scale before and after the injection.

Data Collection Tools Individual Identification Form: Participants' demographic characteristics and injection history.

Injection Fear Scale: 14-item Likert-type scale, 1-5 point range. Visual Analog Scale (VAS): Measurement of pain level after injection using a 0-10 cm line.

Expected Results/Significance The study is expected to determine and compare the effectiveness of ShotBlocker and the Helfer Technique in reducing injection-related pain and fear. The results have the potential to support the use of nonpharmacological methods in clinical practice, thereby increasing patient comfort, ensuring treatment compliance, and improving the quality of nursing care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years.
* Patients diagnosed with breast cancer.
* Requirement of intramuscular (IM) injection of premenopausal or postmenopausal hormonal medications as part of their prescribed treatment.
* Cognitive competence to provide informed consent for the injection procedure. Intact skin integrity and normal sensory perception at the injection site (gluteal region).

Exclusion Criteria:

* History of chronic pain disorders, neuropathic pain syndrome, or any disease requiring regular analgesic use.
* Presence of neurological or cognitive disorders that may alter pain or fear perception.
* Use of analgesics within the last 24 hours (or a specific timeframe relevant to your study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pain Level | Immediately after injection
  Pain will be measured using the Visual Analog Scale (VAS) immediately after intramuscular hormone injection in premenopausal and postmenopausal breast cancer patients. Higher scores indicate higher pain levels.
Injection Fear Scale | The scale will be administered twice: immediately before the injection (baseline) and immediately after the injection.
  The scale developed by Yıldız and Çiftçi (2023) will be used to assess the fear levels of participants regarding the injection procedure. The scale consists of 14 items, rated on a 5-point Likert scale (1 = No fear, 5 = Extreme fear). The total score is calculated as the mean of the item scores, ranging from a minimum of 1 to a maximum of 5. Higher scores indicate higher levels of injection-related fear. The Cronbach's alpha coefficient of the scale was reported as 0.92 in the original study.

CONTACTS AND LOCATIONS:
Locations (1):
- Batman Training and Research Hospital, Batman, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect the privacy and confidentiality of the study participants. The informed consent and ethical approval obtained for this study do not cover the public sharing of raw individual-level data with third parties.

REFERENCES:
- [Background] Yaray O, Akesen B, Ocaklioglu G, Aydinli U. Validation of the Turkish version of the visual analog scale spine score in patients with spinal fractures. Acta Orthop Traumatol Turc. 2011;45(5):353-8. doi: 10.3944/AOTT.2011.2528. PMID 22033000
- [Background] Agac E, Gunes UY. Effect on pain of changing the needle prior to administering medicine intramuscularly: a randomized controlled trial. J Adv Nurs. 2011 Mar;67(3):563-8. doi: 10.1111/j.1365-2648.2010.05513.x. Epub 2010 Dec 28. PMID 21198801
- [Background] Cocoman A, Murray J. Intramuscular injections: a review of best practice for mental health nurses. J Psychiatr Ment Health Nurs. 2008 Jun;15(5):424-34. doi: 10.1111/j.1365-2850.2007.01236.x. PMID 18454829
- [Background] Malkin B. Are techniques used for intramuscular injection based on research evidence? Nurs Times. 2008 Dec 16-2009 Jan 12;104(50-51):48-51. PMID 19165987
- [Background] Small SP. Preventing sciatic nerve injury from intramuscular injections: literature review. J Adv Nurs. 2004 Aug;47(3):287-96. doi: 10.1111/j.1365-2648.2004.03092.x. PMID 15238123
- [Background] Ordu Y, Polat HT, Kucukceran K. Effects of cold needle and ShotBlocker applied in the emergency department on pain and satisfaction in intramuscular injection pain: A randomized controlled trial. Australas Emerg Care. 2025 Sep;28(3):157-162. doi: 10.1016/j.auec.2025.02.001. Epub 2025 Feb 8. PMID 39924365
- [Background] Savci C, Ozkan B, Aciksari K, Solakoglu GA. Effectiveness of Two Different Methods on the Perceived Pain and Satisfaction During Intramuscular Antibiotic Injection: ShotBlocker and Local Vibration. Clin Nurs Res. 2022 Jun;31(5):812-819. doi: 10.1177/10547738211051877. Epub 2021 Oct 11. PMID 34628979